CLINICAL TRIAL: NCT05775458
Title: Role of Glutamate-mediate Excitotoxicity in Invasion and Progression Processes of Glioblastoma Multiforme
Brief Title: Glutamate Excitotoxicity and Its Role in Glioblastoma Biology
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Pietro Mortini, MD, Prof., Head of department, IRCCS San Raffaele
Other Study IDs: NCH02-2020
Record Dates: First submitted 2021-03-02; First posted 2023-03-20 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Brain Tumor, Primary
Keywords: Brain tumor; Glutamate
MeSH Terms: conditions — Brain Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and CSF samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult neurosurgical patients: Adult neurosurgical patients with a brain lesion suspected for GBM, candidate to gross total tumor resection (GTR), followed by radiotherapy and chemotherapy (concomitant and adjuvant).
  Interventions: Diagnostic Test: Blood, CSF and tumor samples

INTERVENTIONS:
Diagnostic Test: Blood, CSF and tumor samples — Blood, CSF and brain tissue sampling of Glu and Glu regulatory proteins.

SUMMARY:
Gliomas are the most frequent type of primary brain tumors in adults; among them glioblastoma multiforme (GBM) is the most malignant, being associated with the worst prognosis. Glutamate (Glu) is an aminoacid, responsible for essential functions in the Central Nervous System (CNS), acting both as metabolite and neurotransmitter. It is essential for regulating cellular metabolism and developmental synaptogenesis, cellular migration, differentiation and death. Recent scientific evidences have demonstrated alteration in Glu synthesis and signaling being directly involved in GBM growth and invasion

DETAILED DESCRIPTION:
Glu and its scavenger's levels are measurable both in serum and in the cerebral-spinal fluid (CSF), thus making them ideal markers for tumor aggressiveness and disease activity as well as a potential target for new therapeutic approaches.

Serum and CSF levels of glutamic oxaloacetic transaminase (GOT1), Glutamate Pyruvate Transaminase (GPT) and glutamate and aspartate levels of a total of 40 patients will be collected.

Molecular biology analyses will be conducted and oncological and imaging data will be collected during follow-up in patients enrolled in the present studies. MRI imaging as well as blood sampling will be performed at definite timepoints (baseline and 3, 6 and 9 months follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a brain lesion suspected for GBM, candidate to gross total tumor resection (GTR), followed by radiotherapy and chemotherapy (concomitant and adjuvant).
* Patient able to provide informed consent.

Exclusion Criteria:

* Age < 18 years
* Liver disease
* Severe anemia (Hb <8mg/dl)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a brain lesion suspected for GBM, candidate to gross total tumor resection (GTR), followed by radiotherapy and chemotherapy (concomitant and adjuvant).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Baseline characterization of Glutamate scavengers (Glu-sca) levels in serum | Baseline (before surgery)
  Serum GOT1 (UI/ml), GPT (UI/ml)
Baseline characterization of Glutamate (Glu) levels in serum | Baseline (before surgery)
  Serum Glutamate (μM/L)
Time changes in Glutamate scavengers (Glu-sca) levels in serum | At 3, 6, 9 months following surgery
  Serum GOT1 (UI/ml), GPT (UI/ml)
Time changes in Glutamate (Glu) levels in serum | At 3, 6, 9 months following surgery
  Serum Glutamate (μM/L)

SECONDARY OUTCOMES:
Characterization of Glutamate scavengers (Glu-sca) levels in cerebrospinal fluid (CSF) | Baseline (before surgery)
  CSF levels GOT1 (UI/ml), GPT (UI/ml)
Characterization of Glutamate (Glu) levels in cerebrospinal fluid (CSF) | Baseline (before surgery)
  CSF levels Glutamate (μM/L)

OTHER OUTCOMES:
Association between Glutamate metabolism and Glioblastoma molecular signature | Baseline levels of markers
  Association between Glu and Glu-scavengers' levels and molecular patterns of Glioblastoma as described by 2021 WHO classification

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Mortini, MD, Prof., Study Director — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olar A, Aldape KD. Using the molecular classification of glioblastoma to inform personalized treatment. J Pathol. 2014 Jan;232(2):165-77. doi: 10.1002/path.4282. PMID 24114756
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Wang W, Shi G, Ma B, Hao X, Dong X, Zhang B. Chemotherapy for Adults with Malignant Glioma: A Systematic Review and Network Meta-Analysis. Turk Neurosurg. 2017;27(2):174-181. doi: 10.5137/1019-5149.JTN.15462-15.0. PMID 27337236
- [Background] Robert SM, Sontheimer H. Glutamate transporters in the biology of malignant gliomas. Cell Mol Life Sci. 2014 May;71(10):1839-54. doi: 10.1007/s00018-013-1521-z. Epub 2013 Nov 27. PMID 24281762
- [Background] de Groot J, Sontheimer H. Glutamate and the biology of gliomas. Glia. 2011 Aug;59(8):1181-9. doi: 10.1002/glia.21113. Epub 2010 Dec 29. PMID 21192095
- [Background] O'Kane RL, Martinez-Lopez I, DeJoseph MR, Vina JR, Hawkins RA. Na(+)-dependent glutamate transporters (EAAT1, EAAT2, and EAAT3) of the blood-brain barrier. A mechanism for glutamate removal. J Biol Chem. 1999 Nov 5;274(45):31891-5. doi: 10.1074/jbc.274.45.31891. PMID 10542215
- [Background] Ruban A, Biton IE, Markovich A, Mirelman D. MRS of brain metabolite levels demonstrates the ability of scavenging of excess brain glutamate to protect against nerve agent induced seizures. Int J Mol Sci. 2015 Feb 2;16(2):3226-36. doi: 10.3390/ijms16023226. PMID 25648322
- [Background] Teichberg VI, Cohen-Kashi-Malina K, Cooper I, Zlotnik A. Homeostasis of glutamate in brain fluids: an accelerated brain-to-blood efflux of excess glutamate is produced by blood glutamate scavenging and offers protection from neuropathologies. Neuroscience. 2009 Jan 12;158(1):301-8. doi: 10.1016/j.neuroscience.2008.02.075. Epub 2008 Mar 18. PMID 18423998
- [Background] Rijpkema M, Schuuring J, van der Meulen Y, van der Graaf M, Bernsen H, Boerman R, van der Kogel A, Heerschap A. Characterization of oligodendrogliomas using short echo time 1H MR spectroscopic imaging. NMR Biomed. 2003 Feb;16(1):12-8. doi: 10.1002/nbm.807. PMID 12577293
- [Background] Roslin M, Henriksson R, Bergstrom P, Ungerstedt U, Bergenheim AT. Baseline levels of glucose metabolites, glutamate and glycerol in malignant glioma assessed by stereotactic microdialysis. J Neurooncol. 2003 Jan;61(2):151-60. doi: 10.1023/a:1022106910017. PMID 12622454
- [Background] Willard SS, Koochekpour S. Glutamate signaling in benign and malignant disorders: current status, future perspectives, and therapeutic implications. Int J Biol Sci. 2013 Aug 9;9(7):728-42. doi: 10.7150/ijbs.6475. eCollection 2013. PMID 23983606
- [Background] Chung WJ, Lyons SA, Nelson GM, Hamza H, Gladson CL, Gillespie GY, Sontheimer H. Inhibition of cystine uptake disrupts the growth of primary brain tumors. J Neurosci. 2005 Aug 3;25(31):7101-10. doi: 10.1523/JNEUROSCI.5258-04.2005. PMID 16079392
- [Background] Ruban A, Berkutzki T, Cooper I, Mohar B, Teichberg VI. Blood glutamate scavengers prolong the survival of rats and mice with brain-implanted gliomas. Invest New Drugs. 2012 Dec;30(6):2226-35. doi: 10.1007/s10637-012-9799-5. PMID 22392507
- [Background] Takano T, Lin JH, Arcuino G, Gao Q, Yang J, Nedergaard M. Glutamate release promotes growth of malignant gliomas. Nat Med. 2001 Sep;7(9):1010-5. doi: 10.1038/nm0901-1010. PMID 11533703
- [Background] Corsi L, Mescola A, Alessandrini A. Glutamate Receptors and Glioblastoma Multiforme: An Old "Route" for New Perspectives. Int J Mol Sci. 2019 Apr 11;20(7):1796. doi: 10.3390/ijms20071796. PMID 30978987
- [Background] Campos F, Rodriguez-Yanez M, Castellanos M, Arias S, Perez-Mato M, Sobrino T, Blanco M, Serena J, Castillo J. Blood levels of glutamate oxaloacetate transaminase are more strongly associated with good outcome in acute ischaemic stroke than glutamate pyruvate transaminase levels. Clin Sci (Lond). 2011 Jul;121(1):11-7. doi: 10.1042/CS20100427. PMID 21265738
- [Background] Campos F, Sobrino T, Ramos-Cabrer P, Castellanos M, Blanco M, Rodriguez-Yanez M, Serena J, Leira R, Castillo J. High blood glutamate oxaloacetate transaminase levels are associated with good functional outcome in acute ischemic stroke. J Cereb Blood Flow Metab. 2011 Jun;31(6):1387-93. doi: 10.1038/jcbfm.2011.4. Epub 2011 Jan 26. PMID 21266984